CLINICAL TRIAL: NCT00815295
Title: Sorafenib and Cetuximab in Recurrent and/or Metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN):a Phase I B/II Trial
Brief Title: Study of Sorafenib/Cetuximab in Head and Neck Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00001516
Record Dates: First submitted 2008-12-26; First posted 2008-12-30 (Estimated); Results first posted 2014-12-08 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Squamous Cell Cancer
Keywords: squamous cell cancer, head and neck
MeSH Terms: conditions — Neoplasms, Squamous Cell | interventions — Sorafenib; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cetuximab + sorafenib (Experimental): Cetuximab will be given at standard approved dose: 400 mg/m2 loading dose followed by 250 mg/m2 weekly. Sorafenib will be given at 200mg/m2 twice daily.
  Interventions: Drug: Sorafenib; Drug: Cetuximab

INTERVENTIONS:
Drug: Sorafenib — Phase 1 - Dose level 1 : Sorafenib will be given 200 mg twice daily oral, Phase 1 - Dose level 2 : Sorafenib will be given 400 mg twice daily oral, Phase 2 : Sorafenib will be given at the maximum tolerated dose from Phase 1
  Other Names: Nexavar
Drug: Cetuximab — Cetuximab will be given at standard approved dose: 400 mg/m2 loading dose followed by 250 mg/m2 weekly.
  Other Names: Erbitux

SUMMARY:
In this Phase I B/II trial, we seek to determine the safety and efficacy of sorafenib with standard dose cetuximab in the treatment of patients with Recurrent and /or Metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN).

DETAILED DESCRIPTION:
This is a non-randomized phase I B/II trial enrolling 43 patients with recurrent and/or metastatic SCCHN who are not candidates for surgical salvage or definitive radiation. Subjects will receive Cetuximab and sorafenib until disease progression. Cetuximab will be given at standard approved dose: 400 mg/m2 loading dose followed by 250 mg/m2 weekly. Sorafenib will be given 200 mg twice daily oral, continuous dosing to the 6 patients in cohort 1. If less than 3 patients experience dose limiting toxicities (DLT) at the 200mg BID dose, then 6 patients will be accrued at the 400mg BID dose level and toxicities will again be examined. Sorafenib will be given 400 mg twice daily oral, continuous dosing to the patients in cohort 2. One cycle equals 28 days. Tumor assessment will be performed every 8 weeks. Treatment continues until disease progression or unacceptable side effects.

Participating subjects will be asked to take part in an optional correlative study to provide previously archived diagnostic or therapeutic tumor samples obtained during the course of their routine medical care for their cancer of the head/neck. The optional tissue repository project is Duke University Health System (DUHS) Institutional Review Board (IRB) approved (eIRB # 11138 / "Tissue Acquisition Protocol for Analysis of Effects of Novel Chemotherapeutic Compounds). Subjects will be asked to sign a separate consent form to participate in the tissue collection study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma of the head and neck
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Age > 18 years old
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
* Adequate bone marrow, liver and renal function as assessed by the following:
* Hemoglobin > 9.0 g/dl
* Absolute neutrophil count (ANC) > 1,500/mm3
* Platelet count > 100,000/mm3
* Total bilirubin < 1.5 times upper limit of normal (ULN)
* Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) < 2.5 times the ULN ( < 5 x ULN for patients with liver involvement)
* Creatinine < 1.5 times ULN
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment
* Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation. Men should use adequate birth control for at least three months after the last administration of sorafenib.
* International normalized ratio (INR) < 1.5 or a Prothrombin Time / Partial thromboplastin time (PT/PTT) within normal limits. Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate. - For patients on warfarin, the INR should be measured prior to initiation of sorafenib and monitored at least weekly, or as defined by the local standard of care, until INR is stable.

Exclusion Criteria:

* Patients must not be candidates for potentially curative complete surgical resection or definitive radiation. (Patients may have received prior chemotherapy as part of definitive chemoradiotherapy and/or for recurrent/metastatic disease)
* Cardiac disease: Congestive heart failure > class II New York Heart Association (NYHA). Patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
* Known brain metastasis. Patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude brain metastasis.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
* Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C.
* Active clinically serious infection > Common Terminology Criteria for Adverse events (CTCAE) Grade 2.
* Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
* Pulmonary hemorrhage/bleeding event > CTCAE Grade 2 (symptomatic and requiring medical intervention) within 4 weeks of first dose of study drug.
* Any other hemorrhage/bleeding event > CTCAE Grade 3 (bleeding requiring blood transfusion or intervention with endoscopy or surgery) within 4 weeks of first dose of study drug.
* Serious non-healing wound, ulcer, or bone fracture.
* Evidence or history of bleeding diathesis or coagulopathy Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug.
* Use of St. John's Wort or rifampin (rifampicin).
* Known or suspected allergy to sorafenib or any agent given in the this trial.
* Any malabsorption problem.
* Previous therapy with cetuximab for the treatment of recurrent and/or metastatic SCCHN. Previous therapy with cetuximab during definitive radiation therapy for locally advanced SCCHN is permitted so long as relapse of SCCHN occurred at least > 6 months (180 days) from the end of cetuximab therapy.
* Previous therapy with sorafenib, sunitinib or another small molecule known to inhibit the vascular endothelial growth factor receptors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Ready, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with recurrent and/or metastatic squamous cell carinoma of the head and neck were enrolled between January 2008 and March 2011. The study was closed prematurely due to poor accrual.
Pre-assignment Details: Three patients were consented to the research study but withdrew consent prior to starting treatment. These patients are not included in the data presented.
Groups:
- Phase 1 - Dose Level 1: Cetuximab was administered at the standard approved dose: 400 mg/m2 loading dose followed by 250 mg/m2 weekly. Sorafenib 200 mg was administered orally twice daily.
- Phase 1 - Dose Level 2: Cetuximab was administered at the standard approved dose: 400 mg/m2 loading dose followed by 250 mg/m2 weekly. Sorafenib 400 mg was administered orally twice daily.
- Phase 2: Cetuximab was administered at the standard approved dose: 400 mg/m2 loading dose followed by 250 mg/m2 weekly. Sorafenib was administered orally twice daily at the MTD from Phase I.
Period: Overall Study
Arm/Group | Phase 1 - Dose Level 1 | Phase 1 - Dose Level 2 | Phase 2
Started | 8 | 8 | 12
Completed | 8 | 7 | 9
Not Completed | 0 | 1 | 3
Not completed — Cetuximab hypersensitivity reaction | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 - Dose Level 1 | Phase 1 - Dose Level 2 | Phase 2 | Total
Number analyzed (Participants) | 8 | 8 | 12 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (7.8) | 61.2 (7.2) | 62.8 (12.3) | 61.0 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 5 | 8
  Male | 6 | 7 | 7 | 20
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 12 | 28

OUTCOME MEASURES:

1. Primary Outcome: Phase 1 - Maximum Tolerated Dose (MTD) of Sorafenib Administered With Cetuximab (400 mg/m2 Loading Dose Followed by 250 mg/m2 Weekly)
Description: The MTD is based upon dose-limiting (DLTs) experienced during Cycle 1 of treatment. The MTD is the maximum dose level at which 0/6 or 1/6 patients experience DLT. Using Common Toxicity Criteria for Adverse EVents (CTCAE) version 3.0, DLTs are defined as any Grade 4 hematologic toxicity, or Grade 3 or 4 non-hematologic toxicity. A DLT will not be considered to have occurred in the case of a grade 3 or 4 allergic reaction due to cetuximab.
Time Frame: Cycle 1 (28 Days)
Population: All patients treated on either dose level 1 or 2 as part of the phase I study.
Measure: Number; unit: mg
Groups:
- Phase 1: Cetuximab was administered at the standard approved dose: 400 mg/m2 loading dose followed by 250 mg/m2 weekly. Sorafenib 200 mg or 400 mg was administered orally twice daily. The dose of sorafenib was escalated from 200 mg to 400 mg in successive 3+3 cohorts of patients to determine the maximum tolerated dose (MTD) of this regimen. The MTD is the maximum dose level at which 0/6 or 1/6 patients experience dose-limiting toxicity (DLT).
Arm/Group | Phase 1
Number analyzed (Participants) | 16
mg | 400

2. Primary Outcome: Tumor Control Rate
Description: The proportion of patients for whom the best overall response is complete response (CR), partial response (PR) or stable disease (SD). A CR occurs when all lesions disappear; whereas, a PR is indicated when there is at least a 30% decrease in the sum of the longest diameters (LD) of the target lesion. A PD (progressive disease) occurs when there is at least a 20% increase in the sum of the LD relative to the smallest sum LD recorded since treatment is initiated. Disease is considered stable if there is no response and no PD. If follow-up assessments are not available, the best overall response is unevaluable.
Time Frame: 1 year
Population: Patients assigned to receive 400 mg of Sorafenib within the phase I or II component of the study are included in the analysis. 4 patients who had a Cetuximab hypersensitivity reaction on day 1 and then terminated treatment are excluded from the analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Subjects Who Received Treatment at the MTD (Phase 1 and 2): Cetuximab was administered at the standard approved dose: 400 mg/m2 loading dose followed by 250 mg/m2 weekly. Sorafenib was administered orally twice daily at 400 mg, the MTD from Phase I.
Arm/Group | Subjects Who Received Treatment at the MTD (Phase 1 and 2)
Number analyzed (Participants) | 16
percentage of participants | 43.8 [19.8 to 70.1]

3. Secondary Outcome: Median Survival
Description: Time in months from the start of study treatment to date of death due to any cause. Median survival was estimated using a Kaplan-Meier curve and is the time point at which 50% of patients remain alive.
Time Frame: 5 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Subjects Who Received Treatment at the MTD (Phase 1 and 2)
Number analyzed (Participants) | 16
months | 9.3 [1.4 to 14.0]

4. Secondary Outcome: Median Progression-Free Survival (PFS)
Description: Time in months from the start of study treatment to the date of first progression (PD) according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria, or death due to any cause. Per RECIST, a PD is indicated when there is at least a 20% increase in the sum of the longest diameters from target lesions relative to the smallest sum recorded since treatment is initiated. Median PFS was estimated using a Kaplan-Meier curve, and is the time at which 50% of patients remain alive without disease progression.
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Subjects Who Received Treatment at the MTD (Phase 1 and 2)
Number analyzed (Participants) | 16
months | 5.6 [1.4 to 7.8]

5. Secondary Outcome: Phase 2 - Mean Change From Baseline in Quality of Life - Functional Assessment of Cancer Therapy - Head and Neck (FACT-H&N)
Description: The outcome measure is the mean change in the Trial Outcome Index (TOI) between baseline and each follow-up assessment measured by the FACT-H&N. The instrument consists of 39 items to assess physical (PWB), social and family (SWB), emotional (EWB), functional well-bing (FWB) and additional head and neck specific concerns (HNCS). Using a 5-point Likert type scale, responses to individual items range from 0 (not at all) to 4 (Very Much) with higher scores indicating better quality of life. The TOI is the sum of PWB (7 items), FWB (7 items) and HNCS scores (12 items). TOI ranges from 0 to 140.
Time Frame: 5 years
Population: QOL data were not consistently collected and can not be analyzed.
Arm/Group | Phase 2
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The adverse events for this study were collected using Common Terminology Criteria for Adverse Events (CTCAE) version 3.0, and have been converted to CTCAE version 4.0 for entry into ClinicalTrials.gov.
Groups:
- Phase 1 - Dose Level 1: Cetuximab was administered at the standard approved dose: 400 mg/m2 loading dose followed by 250 mg/m2 weekly. Sorafenib 200 mg/m2 was administered orally twice daily.
- Phase 1 - Dose Level 2: Cetuximab was administered at the standard approved dose: 400 mg/m2 loading dose followed by 250 mg/m2 weekly. Sorafenib 400 mg/m2 was administered orally twice daily.
Arm/Group | Phase 1 - Dose Level 1 | Phase 1 - Dose Level 2 | Phase 2
Serious Adverse Events (participants affected / at risk) | 1/8 | 1/8 | 5/12
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 - Dose Level 1 (N=8) | Phase 1 - Dose Level 2 (N=8) | Phase 2 (N=12)
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Death NOS (General disorders) | 0 | 0 | 2
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 - Dose Level 1 (N=8) | Phase 1 - Dose Level 2 (N=8) | Phase 2 (N=12)
Anemia (Blood and lymphatic system disorders) | 0 | 2 | 1
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 | 0 | 0
Blurred vision (Eye disorders) | 1 | 0 | 0
Eye disorders - Other, specify (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1
Esophageal pain (Gastrointestinal disorders) | 0 | 1 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 3 | 4 | 1
Nausea (Gastrointestinal disorders) | 2 | 4 | 2
Oral hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 2 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 3 | 0
Edema face (General disorders) | 0 | 1 | 0
Edema limbs (General disorders) | 1 | 1 | 0
Fatigue (General disorders) | 3 | 6 | 3
Fever (General disorders) | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 4 | 2 | 4
Eye infection (Infections and infestations) | 0 | 1 | 0
Tracheostomy site bleeding (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Alkaline phosphatase increased (Investigations) | 0 | 2 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Cholesterol high (Investigations) | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 2
Neutrophil count decreased (Investigations) | 1 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1
Weight loss (Investigations) | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 3 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Dysgeusia (Nervous system disorders) | 2 | 2 | 1
Headache (Nervous system disorders) | 2 | 2 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pharyngeal fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Nail loss (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 4 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Vascular disorders - Other, specify (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No